CLINICAL TRIAL: NCT06961201
Title: A Prospective, Randomized, Parallel-controlled Clinical Study of Nano-crystalline Megestrol Acetate Combined With Standard Treatment Versus Standard Treatment for First-line Extensive-stage Small Cell Lung Cancer (ES-SCLC) in the Cachexia Phase
Brief Title: Nano-crystalline Megestrol Acetate Combined With Standard Treatment Versus Standard Treatment for First-line Extensive-stage Small Cell Lung Cancer in the Cachexia Phase
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Collaborators: West China Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Megaxia ES-SCLC
Record Dates: First submitted 2025-04-29; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-01

CONDITIONS: Extensive-stage Small Cell Lung Cancer (ES-SCLC); The Pre-cachexia or Cachexia Patients Who Have Not Received Systemic Treatment and Are Not Eligible for Curative Therapy
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nano-crystalline Megestrol Acetate Oral Suspension + Standard Therapy (Experimental)
  Interventions: Drug: Nano-crystalline Megestrol Acetate Oral Suspension; Drug: standard treatment
- Standard Therapy (Active Comparator)
  Interventions: Drug: standard treatment

INTERVENTIONS:
Drug: Nano-crystalline Megestrol Acetate Oral Suspension — Nano-crystalline Megestrol Acetate Oral Suspension, with a specification of 125 mg/mL, the study group takes 5 mL orally per day (625 mg/day), and continues medication.
  Arms: Nano-crystalline Megestrol Acetate Oral Suspension + Standard Therapy
Drug: standard treatment — standard treatment

SUMMARY:
This study is a prospective, randomized, parallel-controlled clinical trial, aiming to evaluate the efficacy and safety of nano-crystalline megestrol acetate combined with standard treatment compared to standard treatment alone as first-line therapy for extensive-stage small cell lung cancer (ES-SCLC) in both the pre-cachexia and cachexia phases. Participants enrolled in the study are those with ES-SCLC in the pre-cachexia or cachexia phase who have not received systemic treatment and are not eligible for curative therapy.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2.
* Life expectancy of ≥6 months.
* Histologically or cytologically confirmed extensive-stage small cell lung cancer (ES-SCLC) (according to the Veterans Administration Lung Study Group (VALG) staging system).
* Participants must not have previously received systemic chemotherapy for ES-SCLC. For participants who have previously received adjuvant/neoadjuvant chemotherapy for non-metastatic disease with curative intent or concurrent/sequential chemoradiotherapy for locally advanced disease, they are eligible for this study if disease progression occurs >6 months after the completion of the last treatment.
* Participants who have previously received PD-1/L1 inhibitors in the neoadjuvant setting are allowed to participate in this study after investigator assessment and agreement. Participants who have previously received PD-1/L1 inhibitors in the adjuvant setting or as consolidation therapy after curative chemoradiotherapy are not eligible for this study.
* At least one measurable tumor lesion according to RECIST v1.1.
* Meet the criteria for pre-cachexia or cachexia diagnosis (based on the Fearon diagnostic criteria).

Exclusion Criteria:

* Presence of conditions that may affect gastrointestinal absorption, such as dysphagia, malabsorption, history of gastrectomy, or uncontrollable vomiting; ongoing enteral feeding or parenteral nutrition; or anorexia due to neurological causes, psychiatric conditions, or pain that makes eating difficult.
* Currently taking or planning to take other medications that increase appetite or weight, such as corticosteroids (excluding short-term use of dexamethasone during chemotherapy), androgens, progestogens, thalidomide, olanzapine, anamorelin, or other appetite stimulants.
* Patients with Cushing's syndrome, adrenal or pituitary insufficiency; patients with poorly controlled diabetes mellitus.
* Concurrent enrollment in another clinical trial, unless it is an observational, non-interventional trial or the follow-up period of an interventional study.
* Presence of unresolved toxicities from prior anti-tumor treatments. Unresolved is defined as not having returned to Grade 0 or 1 according to NCI CTCAE Version 5.0 (except for alopecia) or not having returned to the levels specified in the enrollment/exclusion criteria.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects with improved appetite based on A/CS-12 assessment | Week 3
The proportion of subjects with a relative increase in BMI from baseline | Week 12

CONTACTS AND LOCATIONS:
Locations (1):
- West China School of Medicine/West China Hospital of Sichuan University, Chengdu, Sichuan, China